CLINICAL TRIAL: NCT01427959
Title: Tampere Traumatic Head and Brain Injury Study
Acronym: TheBrainS
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Teemu Luoto, Medical Researcher, Tampere University Hospital
Other Study IDs: R10027
Record Dates: First submitted 2011-09-01; First posted 2011-09-02 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. 10ml whole blood
  2. 10ml EDTA-blood x2
Oversight: Data Monitoring Committee: No

SUMMARY:
Tampere Traumatic head and brain injury study is a prospective study aiming to explore neuroradiological, neuropsychological, neurological and biochemical aspects of mild traumatic brain injury (mtbi). The main interest is on factors that effect to the outcome after mtbi. The study is conducted in Tampere University Hospital's emergency department between the 1st of August 2010 and 31st of July 2013.

DETAILED DESCRIPTION:
Aims of the study:

1. To improve clinical assessment of mTBI in the acute phase
2. To assemble better knowledge of diffusion tensor imaging as a diagnostic tool in mTBI
3. To improve neuropsychological evaluation of mTBI Main focus on psychosocial functioning / outcome / correlates E.g. Resilience, PTSD

ELIGIBILITY:
Inclusion Criteria:

* WHO's mtbi criteria
* Inhabitant of Pirkanmaa hospital district
* Age between 18 and 60 years

Exclusion Criteria:

* Detrimental alcohol use
* Drug addiction
* Chronic neurological disease
* Earlier brain injury
* Diagnosed psychiatric disease
* Hearing or sight deficiency
* Native language other than finnish

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample consisting of consecutive mild traumatic brain injury patients metting the enrollment criteria.
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2010-11; Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teemu M. Luoto, M.D., Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland